CLINICAL TRIAL: NCT01660594
Title: Comparison of CT Coronary Artery Calcium Scoring With Traditional Assessment in Patients Presenting to the Rapid Access Chest Pain Clinic With Non-acute Chest Pain and Its Prognostic Value
Brief Title: CT Calcium Scoring in Suspected Stable Angina
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 11/LO/1693
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Disease
Keywords: coronary disease; tomography, x-ray computed; calcium; exercise test
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stable chest pain: All patients presenting with stable chest pain and referred by their general practitioners to the chest pain clinic in the hospital who had CT calcium scoring performed besides standard assessment.
  Interventions: Other: CT calcium scoring

INTERVENTIONS:
Other: CT calcium scoring — CT Calcium scoring was performed in the patients as an imaging test in addition to the traditional assessment on the same day of patients attending the chest pain clinic on the first visit. This was performed with standard protocol and the absolute calcium score was calculated.

SUMMARY:
Patients with stable chest pain presenting to general practitioners in UK are routinely referred to the chest pain clinics in the hospitals. They are assessed by clinical history including risk factors, cardiovascular exam, resting ECG, chest x-ray, and exercise ECG. CT calcium scoring (CTCS) is a technique that is very sensitive in identifying and quantifying calcified atherosclerotic plaques. Recent guidance from the National Institute of Clinical Excellence (NICE, citation 1) proposes the use of CTCS in patients with stable chest pain who have low likelihood of coronary artery disease (CAD). They recommend that patients with low likelihood (10-30%) have a CTCS and if the score is 0, they can be considered to have non-cardiac chest pain. However, there is controversy regarding relationship of absent calcification with significant CAD and its prognostic value.

At our institution, we have been performing CTCS in this patient cohort since 2003. We plan to retrospectively review the usefulness in CTCS in patients with different likelihood for significant CAD, particularly in patients with absent calcium and compare with the traditional assessment. We also plan to follow-up these patients for any myocardial infarction and death from any cause.

DETAILED DESCRIPTION:
The study seeks to determine the usefulness of CT calcium scoring (CTCS) in patients presenting with non-acute chest pain to the rapid access chest pain clinic (RACPC) and compare it with the traditional assessment in predicting significant CAD and outcome with respect to non-fatal MI or death. The clinical, diagnostic, and follow-up data of patients in last 7 years since CTCS has been performed in the hospital would be retrospectively analysed for the purpose.

Background Patients with chest pain (excluding that of sudden onset) are routinely referred by the GPs to the RACPC centres in the hospitals. They are assessed by clinical history including risk factors, cardiovascular exam, resting ECG, chest x-ray, and exercise ECG. At our institution, we have also been performing CTCS in men more than 40 and women more than 50 years of age since 2003. Recent NICE guidance1 recommends that patients with low pre-test probability (10-30%) of significant coronary artery disease (CAD) have a CT calcium scoring scan and if the score is 0, they can be considered to have non-cardiac chest pain. However, there is controversy regarding relationship of absent calcification with significant CAD and its prognostic value.

This study would enable us to compare and determine the value of CTCS in patients with non-acute chest pain in predicting significant CAD and safety of absent coronary artery calcification.

Rationale for Study

1. To determine if CT coronary calcium scoring adds any value to the existing clinical assessment and exercise ECG. This is not well established in patients presenting with non-acute chest pain to the rapid access chest pain clinics.
2. The study would help in determining if absence of calcification on CT can be considered to have low likelihood of significant coronary artery disease and a good cardiovascular outcome over the period of follow-up. Both these issues are currently controversial in the literature in this group of patients.

STUDY OBJECTIVES

Primary Objective To determine the prognostic value of CT coronary calcium scoring in patients with non-acute chest pain for non-fatal MI and death, and compare with traditional assessment including exercise ECG.

Secondary Objectives To determine how CT coronary calcium scoring compare with traditional assessment including exercise ECG in predicting significant coronary artery disease in patients presenting with non-acute chest pain.

METHODOLOGY Design This is a retrospective cross-sectional study involving analysis of patients' clinical, diagnostic, and management data from hospital records and follow-up questionnaires for outcome. The study does not require any new diagnostic, therapeutic, or interventional procedure.

Data of patients who have presented to the chest pain clinic since October 2003 would be collected from hospital records for:

1. Age, sex, type of chest pain, and risk factors. These would be used to calculate the pre-test probability of significant coronary artery disease (CAD) using Duke's score.
2. Results of exercise ECG where performed.
3. Results of CT calcium scoring.
4. Results of other non-invasive investigations such as stress imaging and CT coronary angiography where performed.
5. Results of invasive coronary angiography where performed. Patients with >70% diameter stenosis or those who underwent percutaneous stent insertion (PCI) or bypass surgery would be considered to have significant CAD.

For those patients who do not undergo any PCI or surgery as a result of above evaluation, we will try to find out if they have subsequently suffered any heart attack or died. This would again be performed through hospital records and if not available, through questionnaires send to the patients and/or their GPs as part of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* non-acute chest pain
* those who underwent CT calcium scoring
* availability of all relevant risk factor information

Exclusion Criteria:

* previous coronary disease i.e., myocardial infarction or revascularization

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to our chest pain clinic between October 2003 to March 2010 with stable (non-acute) chest pain and assessed with history, physical examination, cardiovascular risk factors, chest X-ray, 12-lead resting ECG and exercise ECG.
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 7 years

SECONDARY OUTCOMES:
Non-fatal myocardial infarction | 7 years

OTHER OUTCOMES:
Obstructed coronary artery disease | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Harefield Hospital, London, Middlesex, United Kingdom

REFERENCES:
- [Background] Skinner JS, Smeeth L, Kendall JM, Adams PC, Timmis A; Chest Pain Guideline Development Group. NICE guidance. Chest pain of recent onset: assessment and diagnosis of recent onset chest pain or discomfort of suspected cardiac origin. Heart. 2010 Jun;96(12):974-8. doi: 10.1136/hrt.2009.190066. No abstract available. PMID 20538674